CLINICAL TRIAL: NCT03044015
Title: a Primary Care Based Intervention for the Secondary Prevention of Osteoporotic Fractures
Brief Title: Primary Care Based Intervention for the Secondary Prevention of Osteoporotic Fractures
Acronym: APROP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PDMRAL-16
Record Dates: First submitted 2017-01-12; First posted 2017-02-06 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2020-02

CONDITIONS: Osteoporotic Fractures
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): a defined strategy for the identification of OF. To carry out a primary care based intervention about lifestyle, diet and drug prescription, if needed, with an intensive follow-up
  Interventions: Behavioral: community based integrated strategy for secondary prevention of OF
- Control (Active Comparator): Intervention as usual
  Interventions: Behavioral: as usual

INTERVENTIONS:
Behavioral: community based integrated strategy for secondary prevention of OF — Educational programme on pharmacological treatment, diet recommendations, physical activity programme on OF prevention in primary care
  Arms: Intervention
Behavioral: as usual
  Arms: Control

SUMMARY:
BACKGROUND Recent evidence has been published about the effectiveness for the secondary prevention of osteoporotic fractures (OF) of the hospital-based fracture liaison services.

AIM To assess the effectiveness of a primary care based intervention in the secondary prevention of OF.

METHODOLOGY Prospective study of random clusters, defined at the primary-care trust (PCT) level. Total study follow-up 3 years. Sample size 1800 patients.

DESCRIPTION To launch a defined strategy for the identification of OF. To carry out a primary care based intervention about lifestyle, diet and drug prescription, if needed, with an intensive follow-up in the intervention PCT vs treatment as usual in the control branch.

ANALYSIS As the outcome are the new OF, a survival analysis will be done. Risk factors will be analyzed through Cox proportional hazard regression model stratified by age groups.

Outcomes :

* new OF ratio in intervention vs control areas.
* maintenance of the adherence to the pharmacological and non pharmacological interventions proposed
* assessment of cost-effectivity of the intervention

ELIGIBILITY:
Inclusion Criteria:

* Major OF (distal forearm, vertebral, hip, pelvis and humerus
* Caused by a low impact mechanism

Exclusion Criteria:

* High impact mechanism of impact or secondary to other diseases (cancer, Paget disease ...)
* Patients not residing in the area of the targeted primary care practices
* Patients with an invalidating disease (dementia ...)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2017-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with osteoporotic fractures | 24 months

SECONDARY OUTCOMES:
economic cost | 24 months
  We will consider time spent by physicians and nurses, cost of treatment (hospital admissions, drug therapy, rehabilitation)

CONTACTS AND LOCATIONS:
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No